CLINICAL TRIAL: NCT00887757
Title: A Phase 1 Safety and Pharmacokinetic Study of ABT-263 in Combination With Gemzar® (Gemcitabine) in the Treatment of Subjects With Solid Tumors
Brief Title: Safety Study of ABT-263 in Combination With Gemzar (Gemcitabine) in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10-588
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2011-12

CONDITIONS: Solid Tumors
MeSH Terms: interventions — navitoclax; Gemcitabine

ARMS (1):
- gemcitabine +ABT-263 (Experimental)
  Interventions: Drug: ABT-263; Drug: gemcitabine

INTERVENTIONS:
Drug: ABT-263 — 150mg of ABT-263 is taken orally once daily on Days 1-3 and Days 8-10 out of each 21 day cycle.
  325 mg of ABT-263 is taken orally once daily on days 1-3, 8-10, 15-17 out of each 28 day cycle.
  This is a dose escalation study, therefore the dose of ABT-263 will change throughout the study.
  Other Names: navitoclax
Drug: gemcitabine — Gemcitabine 1000 mg/m2 will be given by intravenous infusion on Day 1 and Day 8 of each 21 day cycle. Gemcitabine 1000 mg/m2 will be given by intravenous infusion on days 1, 8 and 15 of each 28 day cycle.
  Other Names: gemzar, gemcitabine

SUMMARY:
This is a Phase 1 open-label study evaluating the safety of navitoclax (ABT-263) when combined with a standard regimen of gemcitabine in approximately 50 subjects with solid tumors and measurable disease.

ELIGIBILITY:
Inclusion Criteria

* Age greater then or equal to 18 years.
* For the 21 and 28-day dose escalation cohorts and the 21-day safety expansion cohort subjects must have histologically and/or cytologically documented cancer for which gemcitabine has been determined to be an appropriate therapy, per the Investigator.
* For the 28-day safety expansion cohort, subjects must have histologically and/or cytologically documented ductal adenocarcinoma or undifferentiated carcinoma of the pancreas for which gemcitabine has been determined to be an appropriate first-line therapy, per the investigator.

Note: If the 28-day dose escalation schedule is deemed intolerable and further dose de-escalation is not explored, the expanded safety cohort will evaluate navitoclax (ABT-263) in combination with gemcitabine in an additional 12 to 15 subjects with histologically ductal adenocarcinoma or undifferentiated carcinoma of the pancreas for which gemcitabine has been determined to be an appropriate first-line therapy with the RPTD and schedule from the 21-day portion of the study.

* Measurable disease by CT or MRI as defined RECIST.
* Subjects with brain metastases must have clinically controlled neurologic symptoms, defined as surgical excision and/or radiation therapy followed by 21 days of stable neurologic function and no evidence of CNS disease progression as determined by CT or MRI within 28 days prior to the 1st dose of study drug.
* ECOG less then or equal to 1.
* Must have adequate bone marrow, renal and hepatic function per local laboratory reference range as follows:

  * Bone marrow:Absolute Neutrophil Count greater then or equal to1500/μL; platelets greater then or equal to 150,000/mm^3; hemoglobin greater then or equal to 9.0 g/dL;
  * Renal function: Serum creatinine less then or equal to 2.0 mg/dL or calculated creatinine clearance greater then or equal to 50 mL/min;
  * Hepatic function and enzymes: AST , ALP and ALT less then or equal to 3.0 × the upper limit of normal (ULN), bilirubin less then or equal to 1.5 × ULN.
  * Subjects with liver metastasis may have AST, ALP, and ALT less then or equal to 5.0 X ULN.
  * Subjects with bone metastasis may have ALP less then or equal to 5.0 × ULN; Coagulation: aPTT and PT not to exceed 1.2 × ULN.
* Female subjects must be surgically sterile, postmenopausal (for at least 1 year), or have negative results for a pregnancy test performed as follows: at Screening via serum sample obtained within 14 days prior to initial study drug administration and prior to dosing via urine sample obtained on Cycle 1 Day 1, if it has been greater then 7 days since obtaining the serum pregnancy test results.
* Female subjects not surgically sterile or postmenopausal (for at least 1 year) and non-vasectomized male subjects must practice at least 1 of the following methods of birth control:

  * total abstinence from sexual intercourse (minimum 1 complete menstrual cycle);
  * vasectomized partner;
  * hormonal contraceptives (oral, parenteral or transdermal) for at least 3 months prior to study drug administration;
  * Double-barrier method (including condoms, contraceptive sponge, diaphragm or vaginal ring with spermicidal jellies or cream).

Exclusion Criteria

* Underlying, predisposing condition of bleeding or currently exhibits signs of bleeding.
* Recent history of thrombocytopenia associated with bleeding w/i 1 year prior to 1st dose of study drug.
* Currently receiving or requires anticoagulation therapy or any drugs or herbal supplements that affect platelet function, w/the exception of low-dose anticoagulation medications that are used to maintain the patency of a central iv catheter.
* Active peptic ulcer disease or other potentially hemorrhagic esophagitis/gastritis.
* Active immune thrombocytopenic purpura, autoimmune hemolytic anemia or a history of being refractory to platelet transfusions (w/i 1 year prior to the 1st dose of study drug).
* Received radio-immunotherapy w/i 6 months prior to 1st dose of study drug.
* Received an antibody therapy or other biologics (with the exception of colony stimulating factors [G-CSF,GM-CSF] or erythropoietin) w/i 28 days prior to 1st dose of study drug.
* Received anti-cancer therapy including chemotherapy, immunotherapy, radiotherapy, hormonal therapy (with the exception of hormones for hypothyroidism, ERT, anti-estrogen analogs, LHRH, GnRH agonists required to suppress serum testosterone levels if on a stable dose for at least 21 days prior to the 1st dose of study drug), or any investigational therapy w/i 14 days prior to the 1st dose of study drug, or has not recovered to less than a grade 2 clinically significant adverse effect(s)/ toxicity(s) of the previous therapy.
* Received steroid therapy for anti-neoplastic intent w/i 7 days prior to the 1st dose of study drug. (Inhaled steroids for asthma, topical steroids, replacement/stress corticosteroids, or corticosteroids taken as premedication for this study will not be considered exclusionary).
* Received aspirin w/i 7 days prior to 1st dose of study drug.
* History of hypersensitivity to gemcitabine.Positive for HIV.
* Significant history of cardiac, renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, or hepatic disease.
* Exhibits evidence of other clinically significant uncontrolled condition; active systemic fungal infection;diagnosis of fever & neutropenia w/i 1 week prior to study drug administration.
* The subject has undergone prior procedures or has active gastrointestinal disease that would result in the inability to adequately absorb an oral medication (e.g., uncontrolled nausea, vomiting, inflammatory disease, bowel obstruction, or a major bowel resection).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Assess the safety profile of ABT-263 in combination with gemcitabine. | Weekly
Study the pharmacokinetic interaction between ABT-263 and gemcitabine. | Weekly
Determine the maximum tolerated dose (MTD) of ABT-263 in combination with gemcitabine. | Weekly

SECONDARY OUTCOMES:
Evaluate safety at the defined recommended Phase 2 dose (RPTD) and schedule in combination with a standard and weekly regimen of gemcitabine. | Bi-monthly
Evaluate preliminary data regarding progression free survival (PFS) | Bi-monthly
Evaluate preliminary data regarding objective response rate (ORR) | Bi-monthly
Evaluate preliminary data regarding time to tumor progression (TTP) | Bi-monthly
Evaluate preliminary data regarding overall survival (OS) | Bi-monthly
Evaluate preliminary data regarding duration of overall response | Bi-monthly
Evaluate preliminary data with Eastern Cooperative Oncology Group (ECOG) performance status | Bi-monthly
Evaluate biomarkers to | Bi-monthly
  Define the relationship between disease states, B-Cell Lymphoma 2 (Bcl-2) family protein expression, and potential response to the proposed therapy navitoclax when added to a standard and weekly regimen of gemcitabine.

CONTACTS AND LOCATIONS:
Overall Officials: Mack Mabry, MD, Study Director — Abbott

REFERENCES:
- [Result] Cleary JM, Lima CM, Hurwitz HI, Montero AJ, Franklin C, Yang J, Graham A, Busman T, Mabry M, Holen K, Shapiro GI, Uronis H. A phase I clinical trial of navitoclax, a targeted high-affinity Bcl-2 family inhibitor, in combination with gemcitabine in patients with solid tumors. Invest New Drugs. 2014 Oct;32(5):937-45. doi: 10.1007/s10637-014-0110-9. Epub 2014 Jun 11. PMID 24916770